CLINICAL TRIAL: NCT00683631
Title: TheraSphere HUD For Treatment of Unresectable HCC
Brief Title: TheraSphere HUD For Treatment of Unresectable Hepatocellular Carcinoma (HCC)
Acronym: TheraSphere
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Collaborators: MDS Pharma Services (Industry)
Responsible Party: Principal Investigator, Robert C. Martin, Professor of Surgery, University of Louisville
Other Study IDs: TheraSphere - 421.03
Record Dates: First submitted 2008-05-16; First posted 2008-05-23 (Estimated); Last update posted 2023-12-18 (Actual); Status verified 2021-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver cancer; liver tumor; HCC; hepatocellular carcinoma; hepatoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- TheraSphere: TheraSphere
  Interventions: Other: TheraSphere HUD

INTERVENTIONS:
Other: TheraSphere HUD — TheraSphere is FDA approved under a Humanitarian Use Device. It is considered a brachytherapy device that delivers intra-arterial radiation therapy using yttrium-90 microspheres directly to liver tumors.
  Other Names: TheraSphere HDE # 980006

SUMMARY:
The purpose of this protocol is to provide access to Therasphere treatment for patients with liver tumors.

DETAILED DESCRIPTION:
Surgical resection of the affected portion of the liver offers the best chance for disease-free survival in patients with primary liver cancer (hepatocellular carcinoma (HCC)). Unfortunately, most of these patients present with disease that is not amenable to surgery (multifocal disease) or have other medical contraindications to surgery (limited hepatic reserve related to advanced cirrhosis or chronic hepatitis). Fewer than 15% of HCC patients are suitable surgical candidates. The objective of treatment with TheraSphere is to selectively administer a potentially lethal dose of radioactive material to cancerous tissue in the liver of patients with HCC. This type of regional therapy may have several advantages over systemically administered treatments and may also be of value as a 'bridging' treatment for HCC patients awaiting a donor organ for liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, of any race or sex, who have histologic proof of primary cancer to the liver, who are able to give informed consent, will be eligible.
* Patients must have an ECOG Performance Status score of greater than or equal to 2, with a life expectancy of > 3 months, non-pregnant with an acceptable contraception in premenopausal women.
* The histopathology confirmation criterion may be waived in patients with a radiographically identifiable liver mass, known laboratory or clinical risk factors for cancer or elevated tumor markers such as AFP (clinical diagnosis).
* Participation in the TheraSphere Registry.

Exclusion Criteria:

* Contraindications to angiography and selective visceral catheterization
* Evidence of potential delivery of greater than 16.5 mCi (30 Gy absorbed dose) of radiation to the lungs
* Evidence of any detectable Tc-99 MAA flow to the stomach or duodenum, after application of established angiographic techniques to stop such flow
* Significant extrahepatic disease representing an imminent life-threatening outcome
* Severe liver dysfunction or pulmonary insufficiency
* Active uncontrolled infection
* Pregnancy
* Refusal to participate in the TheraSphere Registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an observational treatment use protocol that will provide IRB oversight and documentation of the clinical experience of patients undergoing treatment for primary or secondary liver neoplasia using TheraSphere® under an HDE. Participation involves no investigational or research procedures. Patients will be followed for treatment-related adverse experiences for a minimum of 30 days after each treatment. Survival experience will be monitored in accordance with institutional practices.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2004-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Martin, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Hospital / Norton Hospital, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Woodall CE, Scoggins CR, Ellis SF, Tatum CM, Hahl MJ, Ravindra KV, McMasters KM, Martin RC 2nd. Is selective internal radioembolization safe and effective for patients with inoperable hepatocellular carcinoma and venous thrombosis? J Am Coll Surg. 2009 Mar;208(3):375-82. doi: 10.1016/j.jamcollsurg.2008.12.009. PMID 19317999